CLINICAL TRIAL: NCT02580838
Title: The Effects of Early and Late Injection of Botulinum Toxin Type A on Upper Limb Function in Patients With Stroke
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-BR-102-032
Record Dates: First submitted 2015-10-11; First posted 2015-10-20 (Estimated); Last update posted 2022-09-30 (Actual); Status verified 2015-10

CONDITIONS: Stroke
Keywords: Stroke; Spasticity; OnabotulinumtoxinA
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- early OnabotulinumtoxinA group (Experimental): OnabotulinumtoxinA will be injected immediately when spasticity develop in early OnabotulinumtoxinA group.
  Interventions: Drug: OnabotulinumtoxinA
- late OnabotulinumtoxinA group (Active Comparator): OnabotulinumtoxinA will be injected at 6 months after emergence of spasticity in late OnabotulinumtoxinA group.
  Interventions: Drug: OnabotulinumtoxinA
- no OnabotulinumtoxinA group (No Intervention): OnabotulinumtoxinA will not be injected for this group.

INTERVENTIONS:
Drug: OnabotulinumtoxinA — Early OnabotulinumtoxinA group will receive OnabotulinumtoxinA injection when their spasticity develop, late OnabotulinumtoxinA group will have injection at 6 months after emergence of spasticity, the third group will not have OnabotulinumtoxinA intervention.
  Other Names: Botox
  Arms: early OnabotulinumtoxinA group; late OnabotulinumtoxinA group

SUMMARY:
The aim of this study is to determine whether early use of OnabotulinumtoxinA is more effective to improve functional outcomes of upper limb in patients with stroke.

DETAILED DESCRIPTION:
Many patients surviving stroke have significant impairment of function in the affected upper limb due to the development of spasticity. Botulinum toxin type A injection is a powerful treatment option for control of spasticity. In this study, the patients will be randomly assigned into three groups: early OnabotulinumtoxinA group will receive OnabotulinumtoxinA injection when their spasticity develop, late OnabotulinumtoxinA group will have injection at 6 months after emergence of spasticity, the third group will not have OnabotulinumtoxinA intervention. The aim of this randomized controlled study is to evaluate the effects of early and late injection of botulinum toxin type A on upper limb function in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* stroke affecting one body side
* spasticity develops after stroke

Exclusion Criteria:

* musculoskeletal conditions that affected upper limb function prior to stroke
* concurrent use of anti-spasticity medications
* patients with neuromuscular junction or myopathic disorders such as myasthenia gravis or others
* patients with a known allergy to any onabotulinumtoxinA or to any of the excipients of onabotulinumtoxinA (such as human serum albumin)
* patients who are pregnant or may become pregnant at the time of the proposed injection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-08; Primary Completion 2023-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | change from baseline Modified Ashworth Scale at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lin, Principal Investigator — Department of Physical Medicine and Rehabilitation, National Cheng Kung University Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, National Cheng Kung University Hospital, Tainan, Taiwan